CLINICAL TRIAL: NCT01239927
Title: Hartmann vs Resection With Anastomosis and Diverting Stoma for Peritonitis Caused by Perforated Left-sided Colon Diverticulitis: a Multicenter Prospective Randomized Study.
Brief Title: Hartmann vs R/A in Peritonitis by Perforated Diverticulitis
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Ente Ospedaliero Ospedali Galliera (Other)
Responsible Party: Gian Andrea Binda MD, Ente Ospedaliero Ospedali Galliera
Allocation: Randomized | Model: Parallel | Purpose: Treatment
Other Study IDs: PRTHRAPDP
Record Dates: First submitted 2010-11-12; First posted 2010-11-15 (Estimated); Last update posted 2010-11-15 (Estimated); Status verified 2010-07

CONDITIONS: Peritonitis Caused by Perforated Left-sided Colon Diverticulitis
Keywords: diverticulitis; hartmann; anastomosis
MeSH Terms: conditions — Diverticulitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: Primary sigmoid resection with end colostomy (Hartmann)
Procedure: Primary sigmoid resection and immediate anastomosis with diverting stoma (PRA)

SUMMARY:
This prospective randomized trial is to prove the equivalence of primary sigmoid resection with end colostomy(Hartmann)(GROUP A) and primary sigmoid resection and immediate anastomosis with diverting stoma (GROUP B)with regard to morbidity and mortality in patients with peritonitis caused by perforated left-sided colon diverticulitis.

ELIGIBILITY:
Inclusion Criteria:

* Intraoperative demonstrated peritonitis caused by perforated left-sided colon diverticulitis

Exclusion Criteria:

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2000-01; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
30-day mortality and morbidity after emergency surgery | 30-day

SECONDARY OUTCOMES:
30-day mortality and morbidity after elective restoration of intestinal transit | 30 day

CONTACTS AND LOCATIONS:
Overall Officials: Roberto Bergamaschi, MD, Study Chair — Division of Colon & Rectal Surgery State University of New York Stony Brook, New York; Gian Andrea Binda, Study Director — EO Ospedali Galliera, Genova, Italy; Alberto Serventi, Principal Investigator — EO Ospedali Galliera, Genova, Italy
Locations (1):
- Gian Andrea Binda, Genova, Genova, Italy